CLINICAL TRIAL: NCT00784537
Title: Early Salvage With High Dose Chemotherapy and Stem Cell Transplantation in Advanced Stage Hodgkin's Lymphoma Patients With Positive PET After Two Courses of ABVD (PET-2 Positive) and Comparison of RT Versus no RT in PET-2 Negative Patients
Brief Title: High-dose Chemotherapy and Stem Cell Transplantation, in Patients PET-2 Positive, After 2 Courses of ABVD and Comparison of RT Versus no RT in PET-2 Negative Patients
Acronym: HD0801
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIL-HD0801; EudracT Number 2008-002684-14
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's lymphoma; ABVD; FDG-PET (18-Fluoro-deoxy-D-glucose Positron Emission Tomography); Radiotherapy
MeSH Terms: conditions — Hodgkin Disease | interventions — ABVD protocol; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Other): Two courses of ABVD. Early restaging with FDG-PET scan (PET-2)
  The subsequent treatment will be as it follows:
  * PET-2 positive patients will be high-dose salvage treatment;
  * PET-2 negative patients will be treated with four additional courses of ABVD (for a total of six courses).
  The following restaging procedures are planned as it follows:
  * Optional: Whole body CT scan after the fourth course of ABVD; no therapy change will be made according to CT scan.
  * Mandatory: Whole body CT and FDG-PET scans after the sixth course of ABVD (PET-6).
  PET-6 negative patients will be randomized to first arm:
  No radiotherapy.
  Interventions: Drug: ABVD
- Arm B (Other): Two courses of ABVD. Early restaging with FDG-PET scan (PET-2)
  The subsequent treatment will be as it follows:
  * PET-2 positive patients will be high-dose salvage treatment;
  * PET-2 negative patients will be treated with four additional courses of ABVD (for a total of six courses).
  The following restaging procedures are planned as it follows:
  * Optional: Whole body CT scan after the fourth course of ABVD; no therapy change will be made according to CT scan.
  * Mandatory: Whole body CT and FDG-PET scans after the sixth course of ABVD (PET-6).
  PET-6 negative patients will be randomized to second arm:
  Adjuvant radiotherapy (30 Gy) on sites of initial bulky disease.
  Interventions: Drug: ABVD and Radiotherapy

INTERVENTIONS:
Drug: ABVD — ABVD courses are scheduled every 28 days:
  Doxorubicin 25 mg/m2 i.v. day 1 and 15 Bleomycin 10 mg/m2 i.v. day 1 and 15 Vinblastine 6 mg/m2 i.v. day 1 and 15 Dacarbazine 375 mg/m2 i.v. day 1 and 15
  ABVD courses are scheduled every 28 days:
  Doxorubicin 25 mg/m2 i.v. day 1 and 15 Bleomycin 10 mg/m2 i.v. day 1 and 15 Vinblastine 6 mg/m2 i.v. day 1 and 15 Dacarbazine 375 mg/m2 i.v. day 1 and 15
  Randomization to Arm A (Observation)
  Arms: Arm A
Drug: ABVD and Radiotherapy — ABVD courses are scheduled every 28 days:
  Doxorubicin 25 mg/m2 i.v. day 1 and 15 Bleomycin 10 mg/m2 i.v. day 1 and 15 Vinblastine 6 mg/m2 i.v. day 1 and 15 Dacarbazine 375 mg/m2 i.v. day 1 and 15
  Randomization to Arm B, Radiotherapy, in patients in CR, on the area of initial bulky disease (see above for the definition of nodal and/or mediastinal bulk).
  Arms: Arm B

SUMMARY:
The purpose of this study is to define an improvement in patients:

* To evaluate if patients resistant to the initial treatment for residual PET-positive masses after the first two courses of ABVD (PET-2 positive), can be salvaged by early shift to high-dose chemotherapy supported by stem cell rescue
* To analyse if patients achieving early complete response (PET-2 negative), can be spared the adjuvant radiotherapy on areas of initial bulky disease, at the end of the planned six courses of ABVD. To answer this question, PET-2 negative patients will be randomized between radiotherapy versus no radiotherapy at the end of ABVD therapy.

DETAILED DESCRIPTION:
This study is composed by two phases:

1. A phase II multi-centre study evaluating in patients with advanced stage Hodgkin lymphoma the efficacy of an early salvage treatment with high-dose chemotherapy followed by stem cell transplantation in patients FDG-PET positive after two courses of ABVD (PET-2 positive).
2. A phase III randomised study comparing the efficacy of radiotherapy to the areas of initial bulky disease versus no further therapy in PET-2 negative patients in complete remission (PET-6 negative) at the end of six courses of ABVD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin's lymphoma of the classical type (nodular lymphocyte predominance excluded).
* Stage IIB-IV.
* Age 18-70.
* No prior therapy for Hodgkin's lymphoma
* Written informed consent.
* ECOG performance status grades 0-3 (see Appendix E).
* FDG-PET scan before the initiation of treatment.

Exclusion Criteria:

* Prior therapy for Hodgkin's lymphoma.
* Age less than 18 or more than 70.
* Other concomitant or prior malignancies, except basal cell skin carcinoma, or adequately treated carcinoma in situ of the cervix, or any cancer in complete remission for more than 5 years.
* HIV infection.
* Pregnancy or breast-feeding.
* Renal failure (creatinine ≥2 times the normal value), liver failure (AST/ALT or bilirubine ≥ 2.5 times the normal value) or heart failure (NYHA class ≥ 2 or FEV < 45%).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2008-09; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To evaluate if patients resistant to the initial treatment for residual PET-positive masses after the first two courses of ABVD (PET-2 positive), can be salvaged by early shift to high-dose chemotherapy supported by stem cell rescue. | 4 years

SECONDARY OUTCOMES:
To analyse if patients achieving early complete response (PET-2 negative), can be spared the adjuvant radiotherapy on areas of initial bulky disease, at the end of the planned six courses of ABVD. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Levis, MD, Study Director — Ospedale SS. Antonio, Biagio e Cesare Arrigo
Locations (27):
- Italy (27):
  - Centro di riferimento Oncologico Oncologia Medica A, Aviano
  - Università Policlinico di Bari - Divisione di Medicina A, Bari
  - Policlinco Sant'Orsola Isituto di Ematologia ed oncologia Medica, Bologna
  - Sezione di Ematologia Spedali Civili, Brescia
  - Ospedale di Circolo SC Oncologia Medica III, Busto Arsizio
  - Divisione di Ematologia Osp.Businco, Cagliari
  - Policlinico Careggi Cattedra di Ematologia, Florence
  - ASLTO4, Ivrea
  - Osp. Cardinale Panico Divisione di Ematologia Tricase, Lecce
  - Ospedale Niguarda Cà Granda, Milan
  - Università Avogadro Divisione di Ematologia, Novara
  - Ospedale San Francesco UO Ematologia e Centro Trapianti, Nuoro
  - Fondazione Policlinico San Matteo Clinica Ematologica, Pavia
  - Osp. Santa Maria delle Croci UO Ematologia, Ravenna
  - Ospedale Bianchi Melacrino Morelli, Reggio Calabria
  - Osp. degli Infermi Divisione di Oncologia, Rimini
  - Istituto Regina Elena IFO SC Ematologia, Roma
  - Osp.Sant'Eugenio Divisione di Ematologia, Roma
  - Università La Sapienza Dipartimento di Biotecnnologie Cellulari, Roma
  - Istituto Clinico Humanitas Divisione di Oncologia Medica ed Ematologia, Rozzano (MI)
  - AO Universitaria di Sassari, Sassari
  - Policlinico Le Scotte, Siena
  - Struttura Complessa di Onco-Ematologia, Terni
  - IRCC Onco-Ematologia Candiolo, Torino
  - Osp. San Giovanni Battista_Molinette Ematologia 2, Torino
  - Azienda Ospedaliero universitaria di Udine, Udine
  - ASL 14 UO Oncologia, Verbania

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Ricardi U, Levis M, Evangelista A, Gioia DM, Sacchetti GM, Gotti M, Re A, Buglione M, Pavone V, Nardella A, Nassi L, Zanni M, Franzone P, Frezza GP, Pulsoni A, Grapulin L, Santoro A, Rigacci L, Simontacchi G, Tani M, Zaja F, Abruzzese E, Botto B, Zilioli VR, Rota-Scalabrini D, Freilone R, Ciccone G, Filippi AR, Zinzani PL. Role of radiotherapy to bulky sites of advanced Hodgkin lymphoma treated with ABVD: final results of FIL HD0801 trial. Blood Adv. 2021 Nov 9;5(21):4504-4514. doi: 10.1182/bloodadvances.2021005150. PMID 34597375
- [Derived] Zinzani PL, Broccoli A, Gioia DM, Castagnoli A, Ciccone G, Evangelista A, Santoro A, Ricardi U, Bonfichi M, Brusamolino E, Rossi G, Anastasia A, Zaja F, Vitolo U, Pavone V, Pulsoni A, Rigacci L, Gaidano G, Stelitano C, Salvi F, Rusconi C, Tani M, Freilone R, Pregno P, Borsatti E, Sacchetti GM, Argnani L, Levis A. Interim Positron Emission Tomography Response-Adapted Therapy in Advanced-Stage Hodgkin Lymphoma: Final Results of the Phase II Part of the HD0801 Study. J Clin Oncol. 2016 Apr 20;34(12):1376-85. doi: 10.1200/JCO.2015.63.0699. Epub 2016 Feb 16. PMID 26884559